CLINICAL TRIAL: NCT02953223
Title: A Study to Monitor the Use of an Amino Acid-Based Infant Formula
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 15.04.US.HCN
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Cow's Milk Protein Allergy; Eosinophilic Gastrointestinal Disorders; Malabsorption/Maldigestion; Short Bowel Syndrome; Multiple Food Allergies
MeSH Terms: conditions — Milk Hypersensitivity; Eosinophilic Esophagitis; Malabsorption Syndromes; Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Free amino acid infant formula — Patients who will be fed a free amino acid based infant formula

SUMMARY:
To assess the frequency and nature of adverse events in infants fed a free amino acid based infant formula.

DETAILED DESCRIPTION:
Prospective, post-market surveillance program to be conducted in the United States (US). Infant will be invited to enroll by their healthcare provider who recommends the use of a free amino acid based infant formula

ELIGIBILITY:
Inclusion Criteria:

* Infants who use a free amino acid based Infant formula during their first year of life including:

  * Those that are currently consuming the formula at the time of enrollment
  * Those for whom consumption of the formula is planned
* At least one parent/guardian is willing to provide written informed consent form (ICF) for participation in the surveillance program

Exclusion Criteria:

- Infants <37 weeks of corrected gestation age (CGA) at time of enrollment

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The intent of the program is to enroll infants consuming a free amino acid based infant formula identified in the US
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 4 months
  To assess the frequency and nature of adverse events in infants consuming a free amino acid based infant formula

SECONDARY OUTCOMES:
Clinical characteristics | 4 months
  To describe the demographic and clinical characteristics of infants fed a free amino acid based infant formula

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru AraujoTorres, MD, Study Director — Nestle Health Science
Locations (29):
- United States (29):
  - Pediatric Multicare West, Lakeside, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Sutter Institute of Medical Research, Roseville, California
  - Pioneer Clinical Research, Coconut Creek, Florida
  - Children's Center for GI and Nutrition, Hollywood, Florida
  - Childerns Health Center, PA, Homestead, Florida
  - Homestead Medical Clinic, Miami, Florida
  - Next Phase Research, Virginia Gardens, Florida
  - Children's Gastroenterology Speciality, Glenview, Illinois
  - Childrens Health Care, Wheeling, Illinois
  - Springs Medical Research, Owensboro, Kentucky
  - Acadiana Pediatric Gastro and Hep, Lafayette, Louisiana
  - Tulane University Health Sciences Center, Metairie, Louisiana
  - Conduct Clinical Trials, Flushing, New York
  - The Feinstein Institute for Medical Research, Great Neck, New York
  - State University of New York (SUNY), Syracuse, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - UH Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
  - Milestones Pediatric Care, Tulsa, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - Childrens Health Center, PA, Marble Falls, Texas
  - Southwest Children's Research Assoicaites, San Antonio, Texas
  - Dixie Pediatrics, St. George, Utah
  - Multicare Institute for research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No